CLINICAL TRIAL: NCT00677235
Title: A Prospective, Randomized, Concurrently-Controlled Post-Approval Study of the FLAIR Endovascular Stent Graft
Brief Title: Post-Approval Study for the FLAIR Endovascular Stent Graft
Acronym: RENOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPV-07-002
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Stenosis of Vascular Prosthetic Devices, Implants and Grafts
Keywords: Hemodialysis; Vascular Prosthesis; Stenosis; End-stage Renal Disease (ESRD)
MeSH Terms: conditions — Constriction, Pathologic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FLAIR (Experimental): FLAIR Endovascular Stent Graft
  Interventions: Device: FLAIR Endovascular Stent Graft
- PTA Only (Active Comparator): Percutaneous Transluminal Angioplasty
  Interventions: Procedure: PTA

INTERVENTIONS:
Device: FLAIR Endovascular Stent Graft — Treatment of stenoses with primary PTA and placement of the FLAIR Endovascular Stent Graft
  Arms: FLAIR
Procedure: PTA — Treatment of stenoses with PTA only
  Arms: PTA Only

SUMMARY:
The purpose of this study is to confirm the long-term safety and effectiveness of the FLAIR Endovascular Stent Graft for treatment of stenoses at the venous anastomosis of ePTFE or other synthetic arteriovenous (AV) access grafts.

DETAILED DESCRIPTION:
The purpose of the study is to compare efficacy data on subjects randomized to treatment with percutaneous transluminal angioplasty (PTA) and the FLAIR™ Endovascular Stent Graft versus subjects randomized to treatment with PTA only.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be either a male or non-pregnant female greater than or equal to 21 years of age
* Subject is willing to comply with the protocol requirements and can be contacted by telephone
* Subject has a synthetic AV access graft located in an arm that has been implanted for greater than or equal to 30 days and has undergone at least one successful dialysis session prior to the index procedure
* Angiographic evidence (per the institution's standard) is available to indicate that the subject has a stenosis greater than or equal to 50% located at the graft-vein anastomosis of subject's synthetic AV access graft
* The target lesion is estimated to be less than or equal to 7 cm in length (by angiography)
* The entire target lesion is located within 7 cm of the graft-vein anastomosis, as verified by angiography, such that approximately 1 cm of the FLAIR™ Endovascular Stent Graft will extend into non-diseased vein and approximately 1 cm but no more than 2 cm of the FLAIR™ Endovascular Stent Graft will extend into the non-diseased AV graft
* Full expansion of an appropriately sized angioplasty balloon, in the operator's judgment, can be achieved during primary angioplasty
* Graft diameter at the deployment site is between 5 mm and 8 mm as verified by angiography

Exclusion Criteria:

* The subject has a life expectancy of < 25 months.
* The target lesion has had a corresponding thrombosis treated less than or equal to 7 days prior to the index procedure.
* A previously placed stent and/or stent graft located in the treatment area is present. Treatment area includes the entire target lesion and 1 cm of landing zone into both non-diseased AV graft and non-diseased vein.
* The subject has an infected AV access graft or uncontrolled systemic infection.
* The presence of additional lesion(s) in the access circuit less than or equal to 3 cm from the edges of the target lesion that was treated less than or equal to 30 days prior to index procedure.
* The presence of additional lesion(s) in the access circuit > 3 cm from the edges of the primary lesion that are greater than or equal to 30% stenosed. Note: Subjects may be included if the additional lesions(s) can be successfully treated with a final residual stenosis of < 30% prior to the index procedure.
* The location of the target lesion would require that the FLAIR™ Endovascular Stent Graft be deployed fully across the elbow joint (radiographically identified by a combination of the humeroulnar joint and the humeroradial joint).
* The location of the target lesion would require that the FLAIR™ Endovascular Stent Graft cross an angle (between the inflow vein and synthetic AV access graft) that is > 90 degrees.
* The subject has an uncontrolled blood coagulation disorder.
* The subject has a known allergy or sensitivity to contrast media which cannot be adequately pre-medicated.
* The subject has a known hypersensitivity to nickel-titanium.
* Subjects who are currently enrolled or who plan to enroll in other investigations that conflict with follow-up testing or confounds data in this trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ziv Haskal, MD, Principal Investigator — University of Maryland Hospital
Locations (1):
- Access Connections, Bamberg, South Carolina, United States

REFERENCES:
- [Result] Haskal ZJ, Saad TF, Hoggard JG, Cooper RI, Lipkowitz GS, Gerges A, Ross JR, Pflederer TA, Mietling SW. Prospective, Randomized, Concurrently-Controlled Study of a Stent Graft versus Balloon Angioplasty for Treatment of Arteriovenous Access Graft Stenosis: 2-Year Results of the RENOVA Study. J Vasc Interv Radiol. 2016 Aug;27(8):1105-1114.e3. doi: 10.1016/j.jvir.2016.05.019. Epub 2016 Jul 4. PMID 27388566

RESULTS

PARTICIPANT FLOW:
Groups:
- PTA Only: Percutaneous Transluminal Angioplasty (PTA): Treatment of stenoses with PTA only
Period: Overall Study
Arm/Group | FLAIR | PTA Only
Started | 138 | 132
Completed | 97 | 94
Not Completed | 41 | 38
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 37 | 36
Not completed — Adverse Experience | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects with hemodynamically significant stenosis fifty percent, clinical evidence of graft dysfunction (without thrombotic occlusion) at the synthetic AV access graft anastomosis, and who were selected from the Investigator's general subject population were eligible for participation in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | FLAIR | PTA Only | Total
Number analyzed (Participants) | 138 | 132 | 270
Age, Continuous [Median (Full Range); unit: years] | 64 [26 to 89] | 63 [24 to 88] | 63.5 [24 to 89]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 69 | 134
  >=65 years | 73 | 63 | 136
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 86 | 173
  Male | 51 | 46 | 97
Region of Enrollment [Number; unit: participants]
  United States | 138 | 132 | 270

OUTCOME MEASURES:

1. Primary Outcome: ACPP Was Defined as the Interval Following the Index Procedure Until the Next Access Thrombosis or Reintervention.
Description: To demonstrate that the post intervention Access Circuit Primary Patency (ACPP) of FLAIR™ is superior to that of PTA at 12 months post study procedure.
Time Frame: 12 months
Population: All patients who were enrolled in the study were included in the analysis in the treatment group to which they were randomized, regardless of the intervention that they actually incurred (an intent-to-treat analysis).
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
proportion of participants | 0.240 [0.165 to 0.315] | 0.110 [0.054 to 0.167]

2. Primary Outcome: The Index of Patency Function (IPF) [the Average Number of Months Between Interventions] of FLAIR™ is Not Inferior to That of PTA at 12 Months Post Study Procedure.
Description: The IPF is summarized was defined as the time from the index study procedure to complete graft abandonment divided by the number of visits for a reintervention performed on the arteriovenous (AV) access circuit in order to maintain vascular access for hemodialysis.
Time Frame: 12 months
Population: All patients who were enrolled in the study will participate in the analysis in the treatment group to which they were randomized, regardless of the intervention that they actually incurred (an intent-to-treat analysis).Blackwelder t-test testing non-inferiority of the FLAIR® group to that of PTA.
Measure: Least Squares Mean (Standard Deviation); unit: Months/intervention
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
Months/intervention | 5.2 (4.08) | 4.4 (3.51)

3. Primary Outcome: The Number of Participants With Device and/or Procedure Related Adverse Events at 12 Months Post Study Procedure.
Time Frame: 12 months
Measure: Number; unit: Number of Participants with Device and/o
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 128 | 130
Number of Participants with Device and/o | 128 | 130

4. Secondary Outcome: To Assess the Number of Re-interventions to the Access Circuit Until Graft Abandonment or Through 12 Months Post-index Procedure
Description: The estimated number of re-interventions to the access circuit until graft abandonment or through 12 months post-index procedure was a secondary endpoint without hypothesis testing and is therefore summarized descriptively.
Time Frame: Patient Follow-Up
Measure: Mean (Standard Deviation); unit: reinterventions
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
reinterventions | 1.9 (2.18) | 2.4 (2.31)

5. Secondary Outcome: Post-Intervention Assisted Primary Patency at 12 Months
Description: Postintervention assisted primary patency (PAPP) was defined as the interval after the index/study procedure until access thrombosis or a surgical intervention that excluded the treated lesion from the access circuit.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
proportion of participants | 0.497 [0.410 to 0.584] | 0.563 [0.474 to 0.653]

6. Secondary Outcome: Post-intervention Secondary Patency (PSP) at 12 Months
Description: Postintervention secondary patency [PSP; referred to as Access Circuit Cumulative Patency (ACCP) in the pivotal trial] was the interval following the treatment procedure until the access circuit was surgically declotted, revised, or abandoned because of inability to treat the original stenosis.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
proportion of participants | 0.653 [0.569 to 0.736] | 0.710 [0.629 to 0.792]

7. Secondary Outcome: Procedural Success
Description: Procedural success was a secondary endpoint without hypothesis testing and is therefore summarized descriptively. Procedural success is defined as anatomic success and at least one indicator of hemodynamic or clinical success.
Time Frame: Patient Follow-Up
Measure: Number; unit: Percentage of Participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
Percentage of Participants | 81.2 | 75.0

8. Secondary Outcome: Analysis of Proportion of Serious Adverse Events Classified as Device and/or Procedure-Related Through 30 Days Post-Procedure
Description: The incidence of device-related and procedure-related serious adverse events (SAEs) from the index procedure through 30 days post procedure is summarized. The purpose of this analysis was to assess the effectiveness of the Bard Peripheral Vascular (BPV) clinician training program.
Time Frame: Patient Follow-Up
Measure: Number; unit: events
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
events | 2 | 0

9. Secondary Outcome: Demonstrate Non-inferiority of FLAIR Safety in Terms of Serious Adverse Events at 12 Months
Description: Serious Adverse Events at 12 months are reported for all 270 subjects.
Time Frame: 12 months
Measure: Number; unit: percentage of participants with serious
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
percentage of participants with serious | 60.9 | 65.9
Statistical Analysis 1: Comparison: FLAIR vs PTA Only; Test type: Superiority or Other; p = 0.449, Fisher Exact

10. Secondary Outcome: Access Circuit Primary Patency (ACCP) at 24 Months Procedure Until the Next Access Thrombosis or Reintervention.
Description: Access Circuit Primary Patency (ACPP) was defined as the interval following the index procedure until the next access thrombosis or reintervention at 24 months.
Time Frame: 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
proportion of participants | 0.095 [0.029 to 0.162] | 0.055 [0.013 to 0.097]

11. Secondary Outcome: To Estimate Safety at 24 Months.
Description: To estimate the percentage of participants without safety issues through 24 months.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
percentage of participants | 10.9 | 3

12. Secondary Outcome: Post-Intervention Assisted Primary Patency at 24 Months
Description: as for outcome 5
Time Frame: 24 month follow up
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
proportion of participants | 0.384 [0.282 to 0.486] | 0.406 [0.312 to 0.500]

13. Secondary Outcome: Post-intervention Secondary Patency at 24 Months
Description: as for outcome 6
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
proportion of participants | 0.518 [0.410 to 0.626] | 0.574 [0.481 to 0.668]

14. Secondary Outcome: Index of Patency Function (IPF) [the Average Number of Months Between Interventions] Rates of FLAIR™ and PTA at at 24 Months.
Description: The IPF is summarized was defined as the time from the index study procedure to complete graft abandonment divided by the number of visits for a reintervention performed on the AV access circuit in order to maintain vascular access for hemodialysis.
Time Frame: 24 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: Months/intervention
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
Months/intervention | 7.1 (7.04) | 5.3 (5.22)

15. Secondary Outcome: Post-Intervention Assisted Primary Patency at 6 Months
Description: as for outcome 5
Time Frame: 6 month follow up
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
proportion of participants | 0.596 [0.512 to 0.681] | 0.656 [0.573 to 0.740]

16. Secondary Outcome: Post-intervention Secondary Patency at 6 Months
Description: as for outcome 6
Time Frame: 6 month follow-up
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
proportion of participants | 0.748 [0.673 to 0.822] | 0.793 [0.722 to 0.864]

17. Post Hoc Outcome: Treatment Area Primary Patency (TAPP) at 12 Months.
Description: TAPP is defined as patency (open to blood flow) after the study index procedure until reintervention in the treatment area (within 5mm proximal or 5mm distal to the study device or index balloon angioplasty treated area), or thrombotic occlusion that involved the treatment area.
Time Frame: 12 months follow up
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
proportion of participants | 0.476 [0.389 to 0.564] | 0.248 [0.170 to 0.325]

18. Post Hoc Outcome: Treatment Area Primary Patency (TAPP) at 24 Months.
Description: as for outcome 17
Time Frame: 24 months follow-up
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLAIR | PTA Only
Number analyzed (Participants) | 138 | 132
proportion of participants | 0.269 [0.177 to 0.360] | 0.135 [0.068 to 0.202]

ADVERSE EVENTS:
Time Frame: From Index Procedure through 24 months of follow-up.
Arm/Group | FLAIR | PTA Only
Serious Adverse Events (participants affected / at risk) | 84/138 | 87/132
Other Adverse Events (participants affected / at risk) | 128/138 | 127/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLAIR (N=138) | PTA Only (N=132)
Cerebrovascular accident (Cardiac disorders) | 2 (2) | 5 (5)
Congestive heart failure (Cardiac disorders) | 5 (5) | 5 (5)
hemotoma (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 6 (6) | 7 (7)
Infection (Infections and infestations) | 32 (32) | 33 (33)
Pain (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Pseudoaneurysm (Vascular disorders) | 2 (2) | 1 (1)
Significant arm or hand edema (Vascular disorders) | 0 (0) | 1 (1)
Stenosis requiring intervention (Vascular disorders) | 5 (5) | 6 (6)
Thrombotic occlusion (Vascular disorders) | 13 (13) | 3 (3)
Other (Vascular disorders) | 69 (69) | 69 (69)
Perforation (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLAIR (N=138) | PTA Only (N=132)
Cerebrovascular Accident (Vascular disorders) | 0 (0) | 1 (1)
Congestive heart failure (Vascular disorders) | 4 (4) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 3 (3) | 1 (1)
Hemorrhage (Vascular disorders) | 4 (4) | 3 (3)
Hemorrhage (Vascular disorders) | 9 (9) | 8 (8)
Infection (Infections and infestations) | 10 (10) | 4 (4)
Pseudoaneurysm (Vascular disorders) | 7 (7) | 15 (15)
Significant arm or hand edema (Vascular disorders) | 3 (3) | 2 (2)
Steal syndrome (Vascular disorders) | 6 (6) | 3 (3)
Stenosis requiring intervention (Vascular disorders) | 82 (82) | 103 (103)
Thrombotic occlusion (Vascular disorders) | 47 (47) | 45 (45)
Vessel rupture (Vascular disorders) | 2 (2) | 2 (2)
Other (Vascular disorders) | 13 (13) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less